CLINICAL TRIAL: NCT04103775
Title: Mechanisms of Cognitive Change
Acronym: CTCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and intervention halted due to Covid-19 pandemic.
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Michael L Thomas, Assistant Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-8509H
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Remediation (Experimental): Cognitive Remediation comprises of six exercises supplied by BrainHQ by Posit Science Corporation: Sound Sweeps (targets auditory processing speed): Two successive frequency-modulated tone sweeps are presented and participants indicate whether the frequency increased or decreased within each tone: Fine Tuning (targets auditory perception and processing speed): Participants indicate which one of two confusable syllables were presented; Syllable Stacks (targets auditory memory); Users report the order of presented syllables in a serial memory span task; Memory Grid (targets auditory memory); Participants match identical cards representing syllables; To do List Training (targets auditory memory): Participants see a g rid of everyday items (e.g., plant, carrots, shovel) and select the items in accordance with spoken instructions; Rhythm Recall (target auditory memory): Participants recreate auditory melodies
  Interventions: Behavioral: Cognitive Remediation
- Active Control (Active Comparator): Active Control Comprises six exercises also supplied by Post Science Corporation: A Maze Race, Reversi, Bricks Breaking Hex, Word Search II, Bricks Squasher II, and CircloO. These are all common computer games freely offered online.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Cognitive Remediation — See Cognitive Remediation Arm description.
  Arms: Cognitive Remediation
Behavioral: Active Control — See Active Control Arm description.
  Arms: Active Control

SUMMARY:
This study will determine whether targeted cognitive training, a low-cost and low-risk commercial cognitive remediation therapy, directly impacts therapeutic targets as well as secondary outcomes in college undergraduates. The active intervention will be compared to an active control condition (computer games). Participants will also attend CSU TILT (The Institute for Teaching and Learning) Academic Workshops.

DETAILED DESCRIPTION:
The primary goal of this project is to investigate whether commercial cognitive remediation therapy improves cognitive functioning in college undergraduates. The secondary goal is to investigate neurophysiological, cognitive, and psychosocial mechanisms of change. The investigators will compare cognitive remediation therapy to computer games. The active control condition will allow the investigators to determine whether targeted cognitive training, as an adjunct to academic skills training provided by CSU TILT, provides significant improvement over computer games alone (which is also thought to provide some value as "brain training"). Participants who agree to enroll in the study will be randomized to one of two intervention arms: cognitive remediation (CR) or active control (AC). In the CR arm, participants will complete 20 hours of targeted cognitive training, in 30-min session, 5 days per week, over 8 weeks. The AC Arm will follow the same schedule, except that participants will complete video games (e.g., pong). All participants will repeat assessments at randomly determined midpoint, as well as after the 8 weeks of training have been completed.

ELIGIBILITY:
Inclusion Criteria:

* College undergraduate;
* English fluency, and the ability to complete study requirements.

Exclusion Criteria:

* College seniors (i.e., students with more than 89 credits at CSU);
* Students who are concurrently enrolled in another study investigating the efficacy or effectiveness of novel learning or cognitive development techniques (not including tutoring or other existing programs available to CSU undergraduates);
* Participants less than age 15.

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
MATRICS Consensus Cognitive Battery (MCCB) Verbal Learning Subscale Scores | Three time points (1 week pre-randomization, mid-treatment [randomly selected for each participant between the 2nd and 7th week of treatment], and 1 week post-treatment) for all participants.
  Change in MATRICS Consensus Cognitive Battery (MCCB) Verbal Learning Subscale. Demographically corrected T-scores (M = 50; SD = 10; higher better).

SECONDARY OUTCOMES:
Academic Performance | Semester data obtained yearly up to 8 years
  Academic performance will be evaluated using participant grade point average improvement over the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No